CLINICAL TRIAL: NCT07221838
Title: OCTAGON: A Phase 4, Single Arm Study to Investigate Oral Corticosteroid Tapering in Adult Patients With Generalized Myasthenia Gravis Treated With Ravulizumab
Brief Title: A Study to Investigate OCS Tapering in Adult Participants With Generalized Myasthenia Gravis Treated With Ravulizumab
Acronym: OCTAGON
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9281R00005; ALX-MG-502 (Other: Alexion)
Record Dates: First submitted 2025-10-03; First posted 2025-10-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Generalized Myasthenia Gravis; gMG
Keywords: Generalized myasthenia gravis; gMG; Glucocorticoid toxicity; Complement C5 inhibitor; Prednisone reduction; Cortisol monitoring; ravulizumab; corticosteroids; adrenal insufficiency; steroid sparing
MeSH Terms: conditions — Myasthenia Gravis; Adrenal Insufficiency | interventions — ravulizumab; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Corticosteroid Tapering Schedule (Experimental): During the tapering period, participant will follow an Oral Corticosteroid tapering schedule until OCS tapering is complete
  Interventions: Procedure: Oral Corticosteroid Tapering Schedule; Drug: Ravulizumab; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Procedure: Oral Corticosteroid Tapering Schedule — During the tapering period, participant will follow an Oral Corticosteroid tapering schedule as applicable to the participant. The oral corticosteroid (prednisone/prednisolone) is provided as per standard medical care.
Drug: Ravulizumab — Patients being treated with intravenous ravulizumab as part of their standard medical care.
Drug: Prednisone/Prednisolone — Participants will continue with or be switched to prednisone/prednisolone as per standard medical care.

SUMMARY:
This is a prospective, multicenter single arm study designed to evaluate the effectiveness and safety of a predefined oral corticosteroids (OCS) tapering schedule to reduce OCS use in adult participants with acetylcholine receptor positive (AChR+) generalized myasthenia gravis (gMG) being treated with intravenous ravulizumab.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than 18 years and male or female
* Clinical diagnosis of gMG
* Receiving ravulizumab treatment prior to enrollment
* Receipt of OCS therapy equivalent to a daily dose ≥ 7.5 mg of prednisone/prednisolone for ≥ 4 continuous weeks directly preceding enrollment
* A participant of childbearing potential must have a negative highly sensitive pregnancy test (serum or urine, as required by local regulations) taken at Screening before OCS tapering begins.
* Willing to sign informed consent

Exclusion Criteria:

* Concurrent participation in an interventional clinical trial.
* History of chronic hypoadrenalism (ie, Addison's disease).
* Use of concomitant OCS for comorbid conditions other than gMG
* Receipt of a biologic for gMG (e.g., efgartigimod, rozanolixizumab, inebilizumab, rituximab, intravenous immunoglobulin) within 5 half-lives of enrollment
* Pregnant, breastfeeding, or intending to conceive during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2027-08-27 (Estimated); Study Completion 2027-08-27 (Estimated)

PRIMARY OUTCOMES:
Proportion of Adult Participants With gMG Who Either: Discontinue Oral Corticosteroids (OCS) or Reduce Their Daily OCS Dosage ≤ 5 mg/day and Maintain this Status for ≥ 4 Weeks Without Clinical Deterioration of gMG | Up to approximately 32 weeks

SECONDARY OUTCOMES:
Proportion of Adult Participants with gMG Who Discontinue OCS (0 mg/day), Sustained ≥ 4 Weeks Without Clinical Deterioration of gMG | Up to approximately 32 weeks
Percentage Change From Daily OCS Dose (mg/day) at Baseline | Baseline, Up to approximately 32 weeks
Change from Baseline in the Myasthenia Gravis Quality of Life-15 Revised (MG-QoL-15r) Score in Adult Participants with gMG | Baseline, Up to approximately 32 weeks
Change from Baseline in the Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score in Adult Participants with gMG | Baseline, Up to approximately 32 weeks
Cumulative Worsening Score per the Glucocorticoid Toxicity Index - Metabolic Domains (GTI-MD) in Adult Participants with gMG | Baseline up to approximately 32 weeks
Aggregate Improvement Score per the GTI-MD in Adult Participants with gMG | Baseline up to approximately 32 weeks

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Research Site, Chicago, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Neptune City, New Jersey
  - Research Site, Raleigh, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
- Germany (2):
  - Research Site, Bochum
  - Research Site, Essen
- Italy (3):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Rome
- Japan (3):
  - Research Site, Ibaraki
  - Research Site, Kitakyushu-shi
  - Research Site, Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR